CLINICAL TRIAL: NCT01574846
Title: Prospective, Multicentre, Non-interventional (Observational) Study of VANTAS® for the Treatment of Patients With Advanced Prostate Cancer.
Brief Title: Prospective Multicentre Non-interventional Study of VANTAS® for the Treatment of Patients With Advanced Prostate Cancer
Acronym: Vantas
Status: Completed | Type: Observational
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: THE VANTAS STUDY
Record Dates: First submitted 2012-02-15; First posted 2012-04-10 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vantas

SUMMARY:
The aim of this non-interventional (observational) study is to document, in collaboration with established urologists in Scandinavia, experience gained from routine use of Vantas® for the treatment of patients with advanced prostate cancer. In this observational study particular attention will be directed to treatment duration, quality of life and patient and physician acceptance of the medicinal product for long-term therapy. Patient-based measurement parameters such as quality of life and degree of satisfaction will allow registration of information that extends beyond the clinical parameters. The knowledge gathered will enable patient acceptance of long-term therapy to be evaluated. Clinical outcome will also be documented by measuring serum testosterone and prostate specific antigen (PSA) levels.

ELIGIBILITY:
Inclusion Criteria:

* Male patients for whom hormone treatment for advanced prostate cancer is indicated
* Age > 18 years.
* Documented elevated PSA levels.

Exclusion Criteria:

Contraindications for Vantas® (in accordance with Summary of Product Characteristics (SmPC))

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Male patients for whom hormone treatment for advanced prostate cancer is indicated
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2011-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Treatment duration follow-up for each patient. | 1 year

SECONDARY OUTCOMES:
Blood samples | 1 year
  PSA and Testosterone measurement
Quality of Life measurements | 1 year
  EORTC documents

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Björk, MD, Principal Investigator — Urology Dep. Skane University Hospital, Malmoe, Sweden
Locations (1):
- Urology Dep. Skane Univeristy Hospital, Malmo, Sweden